CLINICAL TRIAL: NCT04845490
Title: Comparative Study on the Efficacy of Mitomycin and Lobaplatin in the Treatment of Advanced Colorectal Cancer Patients With Radical Surgery Combined With Hyperthermic Intraperitoneal Chemotherapy
Brief Title: Comparative Study of Mitomycin and Lobaplatin in Advanced Colorectal Cancer Patients With Radical Surgery Combined With Hyperthermic Intraperitoneal Chemotherapy
Acronym: WUHIPEC02
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UHCT-IEC-SOP-016-21-02
Record Dates: First submitted 2021-04-06; First posted 2021-04-15 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2021-04

CONDITIONS: Colorectal Cancer; Chemotherapy Effect; Surgery; Metastasis; Survival
Keywords: advanced colorectal cancer; hyperthermic intraperitoneal chemotherapy; mitomycin; lobaplatin; prognosis
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis | interventions — Mitomycin; lobaplatin

STUDY DESIGN:
Intervention Model Description: We divide patients into 3 groups randomly. drug group 1: Radical Surgery + HIPEC (mitomycin) + mFOLFOX6/XELOX regimen; drug group 2: Radical Surgery + HIPEC (lobaplatin) + mFOLFOX6/XELOX regimen; control group: Radical Surgery + HIPEC (no drug) + mFOLFOX6/XELOX regimen
Who Masked: Participant
Masking Description: the choice of HIPEC drugs is unknown to patients with advanced colorectal cancer, but known to doctors, investigators and outcomes assessors.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Drug group 1 (Experimental): hyperthermic intraperitoneal chemotherapy (HIPEC) (with Mitomycin): Temperature Setting : 43 ± 1.0 ℃. Perfusion time: 60 min. Amount of perfusate: The perfusion fluid is based on the principle of filling the abdominal cavity and unobstructed circulation.
  Choice of perfusate: Normal saline. Drug selection and dose: Mitomycin 30 mg/m2 . Treatment course: 2 times (the first time is after surgery, the second time is 48h after first time).
  Interventions: Drug: Mitomycin
- Drug group 2 (Experimental): hyperthermic intraperitoneal chemotherapy (HIPEC) (with lobaplatin): Temperature Setting : 43 ± 1.0 ℃. Perfusion time: 60 min. Amount of perfusate: The perfusion fluid is based on the principle of filling the abdominal cavity and unobstructed circulation.
  Choice of perfusate: Normal saline. Drug selection and dose: lobaplatin 50 mg/m2 . Treatment course: 2 times (the first time is after surgery, the second time is 48h after first time).
  Interventions: Drug: Lobaplatin
- Control group (No Intervention): hyperthermic intraperitoneal therapy (HIPET) (no drug) : Temperature Setting : 43 ± 1.0 ℃. Perfusion time: 60 min. Amount of perfusate: The perfusion fluid is based on the principle of filling the abdominal cavity and unobstructed circulation.
  Choice of perfusate: Normal saline. Drug selection and dose: no drug. Treatment course: 2 times (the first time is after surgery, the second time is 48h after first time).

INTERVENTIONS:
Drug: Mitomycin — Mitomycin is used as drug for hyperthermic intraperitoneal chemotherapy. Choice of perfusate: Normal saline. Drug selection and dose: Mitomycin 30mg/m2. Treatment course: 2 times (the first time is after surgery, the second time is 48h after first time).
  Arms: Drug group 1
Drug: Lobaplatin — Lobaplatin is used as drug for hyperthermic intraperitoneal chemotherapy. Choice of perfusate: Normal saline. Drug selection and dose: Lobaplatin 50mg/m2. Treatment course: 2 times (the first time is after surgery, the second time is 48h after first time).
  Arms: Drug group 2

SUMMARY:
This study is a prospective, randomized, comparative clinical trial conducted by Wuhan Union Hospital and aim to compare the therapeutic effects of Mitomycin and Lobaplatin in the treatment of advanced colorectal cancer patients with radical surgery combined with hyperthermic intraperitoneal chemotherapy

DETAILED DESCRIPTION:
Hyperthermic intraperitoneal chemotherapy (HIPEC) is traditionally used to treat peritoneal cancer combined with cytoreductive surgery (CRS). Further, there have been more than 20 years for CRS + HIPEC applying in treatment of patients with colorectal cancer peritoneal metastasis. While, to date, the kinds, doses, combinations of HIPEC drugs are not clearly been evaluate a criterion for local advanced colorectal cancer patients. Thus, This study aim to compare the efficacy of Mitomycin and Lobaplatin in the treatment of advanced colorectal cancer patients with radical surgery combined with HIPEC. We plan to recruit 201 patients and divide into 3 groups, 2 drug groups and 1 control group, radomly. all patients with advanced co cancer receive radical surgery + HIPEC + mFOLFOX6/XELOX chemotherapy regimen. the mainly experimental variable is HIPEC drugs and three groups employ Mitomycin, Lobaplatin and none respectively. the endpoints of study include peritoneal metastasis, overall survival, immune status and perioperative safety assessment.

ELIGIBILITY:
Inclusion Criteria:

1. No chemoradiotherapy or other anti-tumor therapy before clinical trial performed;
2. Aged 18-75 years;
3. Male or non-pregnant or lactating women;
4. Pathological diagnosis of colorectal adenocarcinoma;
5. Clinical diagnosis of T3 stage or above without distant metastasis and can be given radical surgery (AJCC Version 8, 2018);
6. Normal function of major organs;
7. Routine blood examinations meeting the following criteria:

   A. HB ≥ 90 g/L; B. ANC ≥ 1.5 x 10 9 /L; C. PLT ≥ 125 × 10 9 /L;
8. Chemistry indexs meeting the following criteria:

   A. TBIL < 1.5ULN; B. ALT and AST < 2.5ULN; ALB > 30 g/L C. serum Cr ≤ 1.25 ULN or endogenous creatinine clearance > 50 ml/min (Cockcroft-Gault formula);
9. ECOG score 0-1;

Exclusion Criteria:

1. A history of other malignant tumors within 5 years;
2. Distant metastasis found during surgery;
3. Allergic to paclitaxel, lobaplatin and other related chemotherapeutic drugs;
4. Suffering from epilepsy or other mental illness, unable to control behavior;
5. Inability to tolerate surgery due to severe cardiac, pulmonary and vascular disease;
6. Pregnant or lactating women.
7. Receiving anti-cancer drug therapy from other clinical trials.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
peritoneal metastasis | 3-year
  peritoneal metastasis-free survival (pRFS)
overall survival | 3-year
  overall survival (OS)

SECONDARY OUTCOMES:
Number of participants with immunosuppression events as assessed by blood immunological indicators | up to 4 weeks
  Before and After Hyperthermic Intraperitoneal Chemotherapy, collect 5mL blood samples of patients for detecting immunological indicators such as CD3, CD4 and CD8 lymphocyte population; Interferon-γ; tumor necrosis factor (TNF)-α; interleukin-2, 4, 8, 10, etc
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | up to 4 weeks
  postoperative adverse events (referring to CTCAE 5.0 [including blood routine, liver and kidney function, patient reaction to HIPEC, adverse events]) was analyzed
The positive rate of cancer cells of participants by exfoliative cytology examination | 1 week
  According to the positive rate of cancer cells measured in exfoliative cytology before and after HIPEC, the difference between the groups is analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Kaixiong Tao, Professor, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology

IPD SHARING:
Plan to Share IPD: Yes
we would like to share IPD to other researchers 1 years after clinical trial finished
Supporting Information: Study Protocol, ICF, CSR
Time Frame: we would like to share IPD to other researchers 1 years after clinical trial finished
Access Criteria: all data should not been used for commercial purpose and other private purpose and only for academic research

REFERENCES:
- [Background] Wisselink DD, Braakhuis LLF, Gallo G, van Grevenstein WMU, van Dieren S, Kok NFM, de Reuver PR, Tanis PJ, de Hingh IHJT. Systematic review of published literature on oxaliplatin and mitomycin C as chemotherapeutic agents for hyperthermic intraperitoneal chemotherapy in patients with peritoneal metastases from colorectal cancer. Crit Rev Oncol Hematol. 2019 Oct;142:119-129. doi: 10.1016/j.critrevonc.2019.06.014. Epub 2019 Jul 9. PMID 31400583
- [Background] Yan TD, Cao CQ, Munkholm-Larsen S. A pharmacological review on intraperitoneal chemotherapy for peritoneal malignancy. World J Gastrointest Oncol. 2010 Feb 15;2(2):109-16. doi: 10.4251/wjgo.v2.i2.109. PMID 21160929
- [Result] Hompes D, Tiek J, Wolthuis A, Fieuws S, Penninckx F, Van Cutsem E, D'Hoore A. HIPEC in T4a colon cancer: a defendable treatment to improve oncologic outcome? Ann Oncol. 2012 Dec;23(12):3123-3129. doi: 10.1093/annonc/mds173. Epub 2012 Jul 25. PMID 22831982
- [Result] Segelman J, Granath F, Holm T, Machado M, Mahteme H, Martling A. Incidence, prevalence and risk factors for peritoneal carcinomatosis from colorectal cancer. Br J Surg. 2012 May;99(5):699-705. doi: 10.1002/bjs.8679. Epub 2012 Jan 27. PMID 22287157
- [Result] Razenberg LG, van Gestel YR, Creemers GJ, Verwaal VJ, Lemmens VE, de Hingh IH. Trends in cytoreductive surgery and hyperthermic intraperitoneal chemotherapy for the treatment of synchronous peritoneal carcinomatosis of colorectal origin in the Netherlands. Eur J Surg Oncol. 2015 Apr;41(4):466-71. doi: 10.1016/j.ejso.2015.01.018. Epub 2015 Jan 29. PMID 25680955
- [Result] Torphy RJ, Stewart C, Sharma P, Halpern AL, Oase K, Herter W, Bartsch C, Friedman C, Del Chiaro M, Schulick RD, Gleisner A, McCarter MD, Ahrendt SA. Dextrose-Containing Carrier Solution for Hyperthermic Intraperitoneal Chemotherapy: Increased Intraoperative Hyperglycemia and Postoperative Complications. Ann Surg Oncol. 2020 Dec;27(13):4874-4882. doi: 10.1245/s10434-020-08330-y. Epub 2020 Apr 19. PMID 32306237

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-26): https://cdn.clinicaltrials.gov/large-docs/90/NCT04845490/Prot_SAP_000.pdf
  • Informed Consent Form (2021-03-26): https://cdn.clinicaltrials.gov/large-docs/90/NCT04845490/ICF_001.pdf